CLINICAL TRIAL: NCT04902937
Title: Association of Adjuvant Radiotherapy of Non-metastatic Breast Carcinoma With Immunomodulation and Circulating Tumor Cell Phenotype in Relation to Patient Age.
Acronym: CETC
Status: Recruiting | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: University Hospital Erlangen (Other); Labor Prof. Pachmann (Unknown)
Responsible Party: Principal Investigator, Matthias Mäurer, Dr. med., University of Jena
Other Study IDs: CETC 002
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Tumor Cell, Circulating
Keywords: Early Stage Breast cancer; Circulating Tumor Cells; Tumor-infiltrating lymphocytes; Radiotherapy; Immunophenotyping
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Radiotherapy, Adjuvant; Mastectomy, Segmental; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Single-cell analyses using qRT-PCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premenopausal patients
  Interventions: Radiation: Adjuvant radiotherapy; Drug: neoadjuvant and adjuvant chemotherapy
- postmenopausal patients
  Interventions: Radiation: Adjuvant radiotherapy; Drug: neoadjuvant and adjuvant chemotherapy

INTERVENTIONS:
Radiation: Adjuvant radiotherapy — Guideline-based therapy of primary non-metastatic early breast carcinoma
  Other Names: breast-conserving therapy
Drug: neoadjuvant and adjuvant chemotherapy — Guideline-based therapy of primary non-metastatic early breast carcinoma

SUMMARY:
In a prospective study, the influence of adjuvant radiotherapy in patients with non-metastatic breast carcinoma on the epithelial tumor cells (CETCs) circulating in the blood and their immunohistochemical characteristics depending on age will be investigated. In addition to a histopathological assignment of the CETCs as cells of the primary tumor, major trigger points of the immune system will be exploratively analyzed.

For this purpose, blood samples are taken from the patients at different time points after tumor resection and during adjuvant radiotherapy. In addition to the detection, isolation and genetic characterization of the CETCs, the determination of immunological biomarkers by immunophenotyping, among other methods, is planned. Furthermore, analyses of tissue from the primary tumor with respect to immunohistochemical features as well as tumor-infiltrating lymphocytes (TILs) are planned. The results will be classified and correlated especially with regard to patient age.

As there are insufficient data available for breast carcinoma regarding radiotherapeutic effects on the immune system depending on patient age, it is of great interest to better understand these molecular biological basics in order to identify potential prognostic biomarkers.

DETAILED DESCRIPTION:
The primary aim of this prospective-explorative phase 0 study is to investigate the influence of adjuvant radiotherapy in patients with non-metastatic breast cancer on the circulating epithelial tumor cells (CETCs) in the peripheral blood and their immunohistochemical characteristics in younger high risk (premenopausal) versus older low risk (postmenopausal) patients. In addition, the immunophenotype will be determined using peripheral venous blood mononuclear cells (PBMCs) at different time points during the course of therapy and correlated with the results of CETC analysis. The aim of the study is to identify prognostic and predictive biomarkers for early stage breast cancer patients. No therapeutic consequences will be derived.

For this purpose, the phenotype and molecular biological profile of CETC will be investigated and compared with the corresponding characteristics of the primary tumor in order to assign the tumor cells detected in the peripheral blood to the primary tumor. In this context, the number of tumor-infiltrating lymphocytes (TILs) will be correlated with circulating tumor cells and immunophenotype.

Another goal is the characterization of individually isolated CETC by RT-PCR. The expression of selected marker genes involved in metastatic processes will be investigated during the course of therapy and compared with that of the primary tumor to identify therapy-associated changes. The in vitro cultivation of so-called tumor spheres and their characterization as a sign of a therapy-resistant phenotype is a secondary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis histologically confirmed invasive breast carcinoma pT1-4 pN0 or pN+ cM0
* curative-intended breast-conserving therapy (BET) ± (neo-) adj. system therapy with subsequent adjuvant radiotherapy of the breast ± lymphatic drainage system planned
* informed consent of the patient

Exclusion Criteria:

* DCIS, Inflammatory breast carcinoma
* Recurrence situation
* Presence of distant metastases
* Second malignancies < 10 years prior to diagnosis of breast carcinoma
* Prior exposure to radiotherapy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Breast cancer
Study Population: Only female patients with non-metastatic breast carcinoma undergoing breast-conserving surgery (± neoadjuvant or adjuvant system therapy) at the Department of Gynecology and Reproductive Medicine Jena followed by adjuvant radiation therapy at the Department of Radiation Oncology and Radiotherapy Jena between June 1, 2021 and June 1, 2023 (recruitment period) will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Age-dependent influence of radiotherapy on circulating epithelial tumor cell counts (CETC) and immunophenotype (PBMC). | observation period 2 years
  Measurement of CETC count / µl blood in the course of therapy and correlation with patient age.
Longitudinal quantification of CETCs as well as immunophenotype at specific time points during the course of therapy. | observation period 2 years
  Measurement of CETC count / µl blood in the course of therapy and correlation with the cell count of detected T and B cells / µl blood.
Comparison of immunohistochemical parameters of the primary tumor with the immunohistochemical and cytological parameters of CETC | observation period 2 years
  Comparison of PD-L1 expression of primary tumor cells with CETC in percent. Comparison of hormone receptor status (estrogen, progesterone) values of primary tumor and CETC in percent.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | observation period 3 years follow up
  Recurrences as a function of time (analysis using Kaplan-Meier curves, log-rank test, and Cox regression).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiooncology, Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: Undecided